CLINICAL TRIAL: NCT00083109
Title: Phase I/II Trial Of Low Dose Suramin (CI-1003, NSC#34936) And 5-Fluorouracil In Patients With Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Fluorouracil and Low-Dose Suramin as Chemosensitization in Treating Patients With Metastatic Renal Cell (Kidney) Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02586; NCI-2012-02586 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCF-6101; NCI-6036; CDR0000363559; CWRU-CASE-1804; IRB 6101 (Other: Cleveland Clinic Foundation); 6036 (Other: CTEP); R01CA093871 (NIH); U01CA062502 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Fluorouracil; dehydroftorafur; Suramin

ARMS (1):
- Treatment (suramin and fluorouracil) (Experimental): PHASE I: Patients receive suramin IV over 30 minutes and fluorouracil IV on days 1, 8, 15, 22, 29, and 36. Cohorts of 3-6 patients receive escalating doses suramin and fluorouracil until the dose level allowing 10-50 uM of suramin into the patient's blood is determined without 2 or more of 6 patients experiencing dose-limiting toxicity.
  PHASE II: Patients receive suramin and fluorouracil (at the dose level determined in phase I) as in phase I.
  In both phases, courses repeat every 8 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Other: Pharmacological Study; Drug: Suramin

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Actino-Hermal; Adrucil; Arumel; Cytosafe; Efudex; Efurix; Fiverocil; Fluoro Uracil; Fluoroplex; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Flurox; Ribofluor; Ro 2-9757; Ro-2-9757; Timazin
Other: Pharmacological Study — Correlative studies
Drug: Suramin — Given IV

SUMMARY:
Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop tumor cells from dividing so they stop growing or die. Suramin may increase the effectiveness of fluorouracil by making tumor cells more sensitive to the drug. This phase I/II trial is studying the side effects and best dose of fluorouracil and the chemosensitizer suramin and to see how well they work in treating patients with metastatic renal cell (kidney) cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose of suramin and fluorouracil that would result in plasma concentrations of suramin between 10-50 uM in patients with metastatic renal cell cancer. (Phase I) II. Determine the objective response rate (complete response and partial response) in patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. Determine the preliminary efficacy of this regimen in these patients. (Phase I) II. Determine the pharmacokinetics of low-dose suramin in these patients. (Phase I) III. Determine the time to tumor progression and progress rate at 3 and 6 months in patients treated with this regimen. (Phase II)

OUTLINE: This is a dose-escalation phase I study followed by a phase II study.

PHASE I: Patients receive suramin IV over 30 minutes and fluorouracil IV on days 1, 8, 15, 22, 29, and 36. Cohorts of 3-6 patients receive escalating doses suramin and fluorouracil until the dose level allowing 10-50 uM of suramin into the patient's blood is determined without 2 or more of 6 patients experiencing dose-limiting toxicity.

PHASE II: Patients receive suramin and fluorouracil (at the dose level determined in phase I) as in phase I.

In both phases, courses repeat every 8 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell cancer

  * Metastatic disease
* Measurable or evaluable disease

  * Measurable disease required for phase II
* No untreated CNS metastasis or CNS metastases progressing ≤ 4 weeks after prior radiotherapy
* Performance status - ECOG 0-1
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* Bilirubin ≤ 1.5 mg/dL
* Creatinine ≤ 1.8 mg/dL
* Calcium ≤ ULN
* No untreated hypercalcemia
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must be surgically sterile or use effective contraception
* No uncontrolled diabetes mellitus
* No known severe hypersensitivity to suramin
* No other concurrent uncontrolled illness
* No active or ongoing infection
* No active autoimmune disease
* No neuropathy ≥ grade 2
* No psychiatric illness or social situation that would preclude study compliance
* No other malignancy within the past 5 years except basal cell skin cancer, carcinoma in situ of the cervix, or localized prostate cancer
* No concurrent filgrastim (G-CSF)
* No more than 2 prior chemotherapy regimens for renal cell cancer (phase II only)
* No concurrent corticosteroid dose more than physiologic replacement levels
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy
* Recovered from prior oncologic or other major surgery
* At least 4 weeks since prior major surgery
* No concurrent surgery
* Recovered from all prior anticancer therapy other than alopecia (chronic toxicity < grade 2)
* At least 4 weeks since prior systemic therapy
* More than 30 days since prior investigational drugs
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-03; Primary Completion 2005-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Dose of suramin to deliver the target plasma concentrations of 10 to 50 uM (Phase I) | Up to 48 hours
Objective response rate (CR + PR) using RECIST criteria (Phase II) | Up to 4 years
  Summary statistics (e.g. means and standard deviations or medians and ranges, or frequency counts) and 95% confidence intervals will be calculated. Graphical models will also be used to summarize the data.

SECONDARY OUTCOMES:
Progression rate (Phase II) | 3 months
  Summary statistics (e.g. means and standard deviations or medians and ranges, or frequency counts) and 95% confidence intervals will be calculated. Graphical models will also be used to summarize the data.
Progression rate (Phase II) | 6 months
  Summary statistics (e.g. means and standard deviations or medians and ranges, or frequency counts) and 95% confidence intervals will be calculated. Graphical models will also be used to summarize the data.
Time to disease progression (Phase II) | Up to 4 years
  Summary statistics (e.g. means and standard deviations or medians and ranges, or frequency counts) and 95% confidence intervals will be calculated. Graphical models will also be used to summarize the data.
Toxicity assessed using NCI CTCAE version 3.0 (Phase II) | Up to 4 years
  Summary statistics (e.g. means and standard deviations or medians and ranges, or frequency counts) and 95% confidence intervals will be calculated. Graphical models will also be used to summarize the data.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Bukowski, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States